CLINICAL TRIAL: NCT01866917
Title: Effectiveness of Transversus Abdominis Plane Block in Reducing Immediate Postoperative Pain in Obese Women After Laparoscopic or Robotic Gynecologic Procedures
Brief Title: Study of TAP and Laparoscopic and Robotic Gynecologic Procedures and Obese Women
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pharmacy stopped dispensing study medication
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-11-397
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Pain
Keywords: Transversis Abdominis Plane Block; obese; robotic surgery; laparoscopic surgery
MeSH Terms: conditions — Pain; Obesity | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP (Experimental): Patients will receive Ropivicaine 0.5% 20cc injectate from a study labeled syringe
  Interventions: Drug: Ropivacaine 0.5% 20cc injectate bilaterally
- Saline (Placebo Comparator): Patients will receive Normal saline 20cc injectate from a study labeled syringe
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine 0.5% 20cc injectate bilaterally
  Arms: TAP
Drug: Placebo
  Other Names: Saline
  Arms: Saline

SUMMARY:
Study the effect of the Transversis Abdominis Plane (TAP) block on pain after surgery for obese women undergoing laparoscopic or robotic gynecologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 30, women undergoing laparoscopic or robotic in-patient procedures

Exclusion Criteria:

* Conversions, non-obese women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ja Hyun Shin, Principal Investigator — Montefiore Medical Center
Locations (1):
- Moses Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Transversus Abdominal Plane: Ropivicaine 0.5% 20cc injectate bilaterally
  Group B
- Saline: Normal saline 20cc injectate bilaterally
  Group A
Period: Overall Study
Arm/Group | Transversus Abdominal Plane | Saline
Started | 17 | 18
Completed | 13 | 12
Not Completed | 4 | 6
Not completed — Pharmacist stopped dispensing treatment | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Transversus Abdominal Plane (Drug B): Ropivicaine 0.5% 20cc injectate bilaterally
- Saline (Drug A): Normal saline 20cc injectate bilaterally
- Total: Total of all reporting groups
Arm/Group | Transversus Abdominal Plane (Drug B) | Saline (Drug A) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Median (Standard Deviation); unit: years] | 45.6 (7.97) | 42.0 (7.97) | 43.8 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Numeric Pain Rating Score (NPRS) 0-10 Scale; (0 is Equivalent to no Pain; 10 is Equivalent to the Worst Pain Imaginable)
Description: Pain assessments by verbal numerical pain score (NPS) at 0, 1 and 2 hours prior to discharge in the Post Anesthesia Care Unit. The 10 point NPS scale ranges from 0-10 with 0 being equivalent to no pain and a value of 10 being equivalent to the worst pain imaginable
Time Frame: 0, 1, and 2 hours
Population: There were 13 participants receiving the Transversus Abdominis Plane TAP (Group B) and 12 participants receiving the placebo Saline (Group A).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Transversus Abdominis Plane (TAP) Group B: Ropivicaine 0.5% 20cc IV bilaterally
- Saline Group A: Normal saline 20cc IV bilaterally
Arm/Group | Transversus Abdominis Plane (TAP) Group B | Saline Group A
Number analyzed (Participants) | 13 | 12
score on a scale
  0 hour | 0 [0 to 8] | 5.5 [0 to 9]
  1 hour | 3 [0 to 8] | 3.5 [0 to 5]
  2 hours | 3 [0 to 6] | 4.5 [0 to 5]
Statistical Analysis 1: Comparison: Transversus Abdominis Plane (TAP) Group B vs Saline Group A; Test type: Superiority; p = .574, Chi-squared

2. Primary Outcome: Postoperative Numeric Pain Score (NPS) 0-10 Scale; (0 is Equivalent to no Pain; 10 is Equivalent to the Worst Pain Imaginable)
Description: Pain assessments by verbal numerical pain score (NPS) at 4, 8, 12 and 24 hours prior to discharge in the Post Anesthesia Care Unit. The 10 point NPS scale ranges from 0-10 with 0 being equivalent to no pain and a value of 10 being equivalent to the worst pain imaginable
Time Frame: 4hrs, 8hrs, 12hrs, and 24hrs.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Transversus Abdominis Plane (TAP) Group B: Ropivicaine 0.5% 20cc injectate bilaterally
  Ropivacaine 0.5% 20cc injectate bilaterally
- Saline Group A: Normal saline 20cc injectate bilaterally
Arm/Group | Transversus Abdominis Plane (TAP) Group B | Saline Group A
Number analyzed (Participants) | 13 | 12
score on a scale
  4 hours | 0 [0 to 7] | 5.5 [0 to 6]
  8 hours | 1 [0 to 5] | 2 [0 to 6]
  12 hours | 2 [0 to 6] | 3 [0 to 5]
  24 hours | 3 [0 to 6] | 1.5 [0 to 7]
Statistical Analysis 1: Comparison: Transversus Abdominis Plane (TAP) Group B vs Saline Group A; TAP has been demonstrated to have a potential role in reducing pain, post-operative opioid requirement, and time to hospital discharge after abdominal hysterectomies and cesarean sections; Test type: Superiority — Statistical analysis performed using SPSS software, version 15 (SPSS Inc., Chicago, IL). Data for quantitative variables reported as a median and interquartile range. The Mann Whitney and chi-square tests were used for the analysis of continuous and categorical variables; p = .825, Chi-squared — Effect size was calculated for the numeric pain rating scale at the immediate post-operative period, 4-hour, 8-hour , 12-hour, and 24-hour time periods as a means to assess post-operative pain control; Interquartile range (IQR) = 3

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Group B (TAP Block); Group A (Saline): The anesthesiologist performing the TAP block will administer an injectate of either normal saline or the TAP block in a study labeled syringe that will be drawn by an OR staff member not involved in the surgery or analysis of study data. The protocol is as follows-- prior to skin incision, under ultrasound guidance, the abdominal wall muscular layers will be identified. A linear 6-13 MHz ultrasound transducer will be used. Once the plane is clearly identified between the internal oblique and transversus abdominal muscles, a 20cc injectate of saline or Ropivacaine 0.5% will be administered bilaterally under direct visualization at the site target using a 2 or 4 inch stimiplex needle depending on the size of the patient.
Arm/Group | Group B (TAP Block) | Group A (Saline)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitations of this study include interim analysis with limited sample size, thus it may result in inadequate power. Early termination due to pharmacist refusal to dispense the experimental Rx (no AEs/SAEs recorded). Only an abstract was written.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes